CLINICAL TRIAL: NCT05069571
Title: Explore the Relationship Between the Percentage of Overspeed of Colonoscopy Withdrawal and the Rate of Adenoma Detection:a Prospective、Multicenter、Observational Study
Brief Title: Endoangel Withdrawal Overspeed Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: EA-21-009
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Endoangel — Collecting the colonoscopy videos and analyzing the correlation between withdrawal overspeed proportion and adenoma detection rate.

SUMMARY:
Exploring the relationship between the percentage of overspeed of colonoscopy withdrawal and the rate of adenoma detection.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are over 18 years old (inclusive);
2. Enteroscopy and related examinations are needed to further clarify the characteristics of digestive tract diseases;
3. Able to read, understand and sign the informed consent form;
4. The researcher believes that the subject can understand the process of the clinical research, is willing and able to complete all the research procedures and follow-up visits, and cooperate with the research procedures.

Exclusion Criteria:

1. Participated in other clinical trials, signed an informed consent form and within the follow-up period of other clinical trials;
2. Abuse of drugs or alcohol or mental disorders in the last 5 years;
3. Women during pregnancy or breastfeeding;
4. Subjects with previous history of bowel surgery;
5. The investigator believes that the subject is not suitable for enteroscopy and related examinations;
6. The investigator believes that the subject is not suitable for high-risk diseases or other special circumstances to participate in clinical trials.
7. Patients with gastrointestinal bleeding;
8. Known or highly suspected allergy to any ingredient of bowel cleansing agent;
9. Restricted activities or any mental or physical condition impairs their ability to drink intestinal cleansing preparations;
10. Known or suspected intestinal obstruction or perforation, toxic megacolon, most colectomy, heart failure (grade III or IV), severe cardiovascular disease, severe liver failure or end, renal insufficiency, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients need to receive the colonoscopy examination.
Sampling Method: Probability Sample
Enrollment: 1210 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 3 months

SECONDARY OUTCOMES:
Proportion of withdrawal overspeed | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided